CLINICAL TRIAL: NCT02787538
Title: Supporting Patient Care With Electronic Resources in the United States (SuPER-US): Effectiveness of an Online Decision Aid for Patients Considering Biologic Therapy for Rheumatoid Arthritis
Brief Title: Supporting Patient Care With Electronic Resources in the United States
Acronym: SuPER-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Arthritis Research Centre of Canada (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Hyon Choi, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015P002116
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Decision Aids; Biologics
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- US-ANSWER-2 decision aid (Experimental): The intervention group will receive simple instructions to access the US-ANSWER-2 decision aid and complete the program on their own computers within two days. At the end of the session, US-ANSWER-2 will produce a one-page summary with the participant's questions, concerns, and preferred medication option.
  Interventions: Behavioral: US-ANSWER-2 decision aid
- Control group (Online medication guide) (Active Comparator): The control group will receive the online medication guide, reflective of usual practice. The online medication guide contains standard information about biologics, including an introduction about biologic options, dosages, and effects.
  Interventions: Behavioral: Control group (Online medication guide)

INTERVENTIONS:
Behavioral: US-ANSWER-2 decision aid — US-ANSWER-2 will consist of: 1) an Information Module that presents effectiveness and side effects of each treatment option, and 2) an interactive Value Clarification Module that guides patients to consider what matter to them the most, and the pros and cons of each treatment option. Within the Information Module, the decision support information (i.e., the benefits and harms of treatment options) will be presented in narrated text, graphics, and a series of animated patient stories demonstrating attributes required for effective communication with doctors and significant others.
  Arms: US-ANSWER-2 decision aid
Behavioral: Control group (Online medication guide) — Standard online medication guide.
  Arms: Control group (Online medication guide)

SUMMARY:
This proof-of-concept randomized trial evaluates the effectiveness of using an online decision aid (US-ANSWER-2) in the decision-making to start or switch biologic therapy in US patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
The proposed project aims to improve the process of making evidence-informed treatment decisions by patients with rheumatoid arthritis (RA) and ultimately empower patient self-management. Current RA treatment emphasizes: 1) the need for early and aggressive treatment, and 2) the use of a treat-to-target approach. However, patients often struggle with treatment decisions, especially when the options have both benefits and risks. To address this challenge, investigators based at Arthritis Research Canada have previously developed an online decision aid called ANSWER-2 (ANimated, Self-serve, WEb-based, Research Tool: Version 2) for RA patients who are considering a biologic, and this tool has been recently adapted for the US healthcare setting (called US-ANSWER-2).

Objectives: 1) To evaluate the effectiveness of US-ANSWER-2 in reducing patients' decisional conflict. 2) To assess the extent to which US-ANSWER-2 improves patients' knowledge about RA medications and confidence in managing their health. 3) To examine the experiences of patients and rheumatologists in using US-ANSWER-2.

The investigators will conduct a proof-of-concept randomized controlled trial with 80 patients with RA. Eligible individuals are those: 1) with a diagnosis of RA from a rheumatologist, 2) whose rheumatologists have recommended initiating a biologic or switching to another biologic, and 3) who have internet access and email. The Intervention Group will receive simple instructions to access the US-ANSWER-2 decision aid and complete the program on their own within two days. At the end of the session, a one-page summary will be produced to help them discuss their questions, concerns, and preferred choices with their health care providers. The Control Group will receive a standard online medication guide, reflective of usual practice. Participants will complete the Decisional Conflict Scale (primary outcome) before and after the intervention (US-ANSWER-2 or standard online medication guide). The following secondary outcome measures will be collected at baseline, Month 1, and Month 2: 1) Medication Education Impact Questionnaire, and 2) Partners in Health Scale. In addition, the use of healthcare resources will be collected at baseline and Month 2, and the use of biologics will be collected at Month 6. All participants and their rheumatologists will be invited to participate in a qualitative interview about their experience with the patient decision aid.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are as follows:

  1. with a diagnosis of RA from a rheumatologist
  2. whose rheumatologists have recommended initiating a biologic or switching to another biologic
  3. who have internet access and email.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) | Change measure (baseline score compared to after using the US-ANSWER-2 intervention at Month 1)
  The Decisional Conflict Scale (short version) measures personal perceptions of uncertainty in choosing options, factors contributing to uncertainty, and effective decision-making. It is one-dimensional and has 10 questions and three response categories (yes/no/unsure) used to compute one score.

SECONDARY OUTCOMES:
Medication Education Impact Questionnaire (MeiQ) | Change measure (baseline score compared to after using the US-ANSWER-2 intervention at Month 1 and at Month 2
  The MeiQ consists of 6 subscales and a total of 29 items. MeiQ was developed and tested in three different samples of patients with rheumatic conditions on their knowledge of medications.
Partners in Health Scale (PHS) | Change measure (baseline score compared to after using the US-ANSWER-2 intervention at Month 1 and at Month 2
  The Partners in Health Scale is an 11-item measure designed to assess self-efficacy, knowledge of RA and treatment, and self-management behaviours such as taking medication appropriately and adopting a healthy lifestyle.
Health Resource Utilization (HRU) Questionnaire | Change measure (baseline score compared to after using the US-ANSWER-2 at Month 2)
  The HRU questionnaire was developed for both self and interviewer administration in people with arthritis and other chronic conditions. It consists of a series of open-ended questions about individuals' visits to health professionals, use of investigative tests, hospital visits, use of medications, purchases of adaptive aids, and estimable productivity loss incurred by the individual and their caregivers due to his/her health.

OTHER OUTCOMES:
Use of biologics | 6 months from baseline
  Patients will be asked whether they started or switched a biologic, and the name, since using the US-ANSWER-2.

CONTACTS AND LOCATIONS:
Overall Officials: Hyon K Choi, MD, DrPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States